CLINICAL TRIAL: NCT04172506
Title: A Multicenter, Open-label, Phase Ib/II Study to Evaluate the Efficacy and Safety of Anti-PD-1 Antibody AK105 in Patients With Selected Advanced Solid Tumors
Brief Title: A Study to Evaluate the Efficacy and Safety of Anti-PD-1 Antibody AK105 in Patients With Selected Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK105-204
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor; Lung Cancer; HCC
Keywords: Anti-PD-1; immunotherapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AK105 (Experimental): AK105 200 mg, every 2 weeks
  Interventions: Drug: AK105

INTERVENTIONS:
Drug: AK105 — Anti-PD-1 antibody

SUMMARY:
This is a multi-center, multi-cohort, open-label, phase Ib/II study to evaluate the efficacy, safety, PK characteristics, immunogenicity and potential biomarkers of AK105 monotherapy in the patients with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Written and signed informed consent.
2. Aged over 18 and less than 75 years at the time of signing the informed consent form, both female and male.
3. ECOG PS is 0-1.
4. The expected survival time is ≥ 3months
5. Histologically or cytologically confirmed selected advanced solid tumor.
6. Subject must have at least one measurable lesion according to RECIST Version1.1.
7. Available archived tumor tissue sample to allow for correlative biomarker studies. In the setting where archival material is unavailable or unsuitable for use, the subject must consent and undergo fresh tumor biopsy.
8. Adequate organ function.
9. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception from Day 1 and for 120 days after the last dose of investigational product.
10. Nonsterilized males who are sexually active with a female partner of childbearing potential must use highly effective method of contraception from Day 1 and for 120 days after the last dose of investigational product.
11. Be willing and able to comply with scheduled visits, treatment regimens, laboratory tests and other requirements for the study.

Exclusion Criteria:

1. Had received experimental drug or used experimental device in the past within 4 weeks prior to the first dose of study drug.
2. Receipt of last radiotherapy or any anti-tumor treatment [chemotherapy, targeted therapy, immunotherapy, Chinese patent drugs with antitumor indications, or immunomodulators or tumor embolization] within 4 weeks prior to the first dose of study drug.
3. Had received any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, etc.), or any other antibody or drug therapy for T cell co-stimulatory or checkpoint pathways (such as ICOS, CD40, CD137, GITR, OX40 antibody or drug), immunocytotherapy, therapeutic antibody, etc.).
4. Toxicity from previous anti-cancer therapy has not been alleviated or resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria.
5. Patients with active, known or suspected autoimmune disease, or a medical history of autoimmune disease, with the exceptions of the following: vitiligo, alopecia, Grave disease, psoriasis or eczema not requiring systemic treatment within the last 2 years, hypothyroidism (caused by autoimmune thyroiditis) only requiring steady doses of hormone replacement therapy and type I diabetes only requiring steady doses of insulin replacement therapy, or completely relieved childhood asthma that requires no intervention in adulthood, or primary diseases that will not relapse unless triggered by external factors.
6. Active or previously recorded inflammatory bowel diseases (e.g. Crohn's disease, ulcerative colitis, or chronic diarrhea).
7. Patients with a condition requiring systemic treatment with either corticosteroid (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration.
8. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
9. Large surgical procedures (defined by researchers as open biopsy, severe trauma, etc.) were performed within 28 days prior to the first dose of study drug.
10. Known history of interstitial lung disease.
11. Patients with untreated chronic hepatitis B or HBV DNA exceeding 1000IU/mL or active hepatitis C. Patients with HCV antibody positive are eligible to participate in the study if the results of HCV RNA test show negative.
12. Patients with active tuberculosis (TB).
13. History of known primary immunodeficiency virus infection or positive HIV testing.
14. Severe infections within 4 weeks prior to the first dose of study drug, including but not limited to complications, sepsis or severe pulmonary infections requiring hospitalization.
15. Patients with meningeal metastasis, spinal cord compression, pia mater disease or active brain metastasis. Patients who meet one of the following requirements may be enrolled: a). No central nervous system metastasis symptoms and signs, such as neurological dysfunction, epilepsy or other central nervous system metastasis before admission. No edema around the lesion found by imaging examination, and no brain metastasis more than 1.5 cm in length. b). Patients with central nervous system metastasis had received treatment and achieved asymptomatic status (e.g. without neurological dysfunction, epilepsy or other typical central nervous system metastasis symptoms and signs)
16. Patients with pleural effusion, pericardial effusion or ascites that could not be controlled stably by repeated drainage or other methods as judged by the investigator.
17. Receipt of live, attenuated vaccination within 30 days prior to the first dose of study treatment, or plan to receive live, attenuated vaccine during the study.
18. Known history of sever hypersensitivity reaction to other monoclonal antibodies.
19. Known history of allergy or hypersensitivity to AK105 or any of its components
20. Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | the time of informed consent signed through 90 days after the last dose of AK105
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Duration of response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Minimum observed concentration (Cmin) of AK105 at steady state | From first dose of AK105 through to 90 days after last dose of AK105
  The endpoints for assessment of PK of AK104 include serum concentrations of AK105 at different timepoints after AK105 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK105 through to 90 days after last dose of AK105
  The immunogenicity of AK105 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Nong Xu, MD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Pang X, Zhong T, Qu T, Chen N, Ma S, He X, Xia D, Wang M, Xia M, Li B. Penpulimab, an Fc-Engineered IgG1 Anti-PD-1 Antibody, With Improved Efficacy and Low Incidence of Immune-Related Adverse Events. Front Immunol. 2022 Jun 27;13:924542. doi: 10.3389/fimmu.2022.924542. eCollection 2022. PMID 35833116
- [Derived] Zheng Y, Mislang ARA, Coward J, Cosman R, Cooper A, Underhill C, Zhu J, Xiong J, Jiang O, Wang H, Xie Y, Zhou Y, Jin X, Li B, Wang ZM, Kwek KY, Xia D, Xia Y, Xu N. Penpulimab, an anti-PD1 IgG1 antibody in the treatment of advanced or metastatic upper gastrointestinal cancers. Cancer Immunol Immunother. 2022 Oct;71(10):2371-2379. doi: 10.1007/s00262-022-03160-1. Epub 2022 Feb 15. PMID 35165764
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10991425/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38412283/